CLINICAL TRIAL: NCT04902885
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Phase 3 Study Evaluating Efficacy, Safety and Pharmacokinetics of Trilaciclib In Extensive-Stage Small Cell Lung Cancer Patients
Brief Title: Phase 3 Study Evaluating Efficacy, Safety and Pharmacokinetics of Trilaciclib In Small Cell Lung Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Collaborators: G1 Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B02B00801-TRILA-301
Record Dates: First submitted 2021-05-08; First posted 2021-05-26 (Actual); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-04

CONDITIONS: Extensive-stage Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — trilaciclib; Carboplatin; Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Part I ( Safety run-in and PK Evaluation); Trilaciclib Group (Active Comparator): 12 patients( 6 patients are first line, 6 patients are second or third line) recieved Trilaciclib(240mg/m^2) plus chemotherapy.
  Interventions: Drug: Trilaciclib, carboplatin, etoposide，or Topotecan
- Part II ( Randomized Double-blind, Placebo-controlled ), Trilaciclib Group (Active Comparator): 41 patients received trilaciclib(240mg/m^2) plus chemotherapy
  Interventions: Drug: Trilaciclib, carboplatin, etoposide，or Topotecan
- Part II ( Randomized Double-blind, Placebo-controlled ), Placebo Group (Placebo Comparator): 42 patients received placebo plus chemotherapy
  Interventions: Drug: placebo, carboplatin, etoposide，or Topotecan

INTERVENTIONS:
Drug: Trilaciclib, carboplatin, etoposide，or Topotecan — Trilaciclib plus carboplatin, etoposide for first line patients ;Trilaciclib plus Topotecan for second or third line patients
  Other Names: Trilaciclib plus chemotherapy
  Arms: Part I ( Safety run-in and PK Evaluation); Trilaciclib Group; Part II ( Randomized Double-blind, Placebo-controlled ), Trilaciclib Group
Drug: placebo, carboplatin, etoposide，or Topotecan — placebo plus carboplatin, etoposide for first line patients ;placebo plus Topotecan for second or third line patients
  Other Names: placebo plus chemotherapy
  Arms: Part II ( Randomized Double-blind, Placebo-controlled ), Placebo Group

SUMMARY:
A Randomized, double-blind, placebo-controlled, multi-center Phase 3 study evaluating efficacy, safety and pharmacokinetics of Trilaciclib In Extensive-Stage Small Cell Lung Cancer Patients Receiving Carboplatin combined with Etoposide or Topotecan The study consists of 2 parts: Part 1: safety run-in and pharmacokinetics evaluation of 12 ES-SCLC patients (6 each for first line and second/third line ES-SCLC patients); Part 2: randomized, double-blind, placebo-controlled efficacy confirmation study of 80 ES-SCLC patients (stratified by first line and second/third line ES-SCLC, ECOG PS [0-1 vs 2] and brain metastases.

The study includes screening period, treatment period, safety follow-up and survival follow-up.

DETAILED DESCRIPTION:
This is a multi-center Phase 3 clinical trial with an open-label single-arm safety run-in and PK evaluation part and a randomized double-blind, placebo controlled part in patients with ES-SCLC to evaluate the safety, efficacy, and pharmacokinetic profile of Trilaciclib based on completed clinical studies abroad.

The study consists of 2 parts. The first part, safety run-in and PK evaluation, enrolled approximately 12 patients with extensive-stage small-cell lung cancer, 6 patients each with 1st line ES-SCLC and 2nd/3rd line ES-SCLC to receive Trilaciclib in combination with carboplatin and etoposide (EC regimen) or with topotecan, and based on evaluable data from Cycle 1, evaluated the safety, tolerability, pharmacokinetics, and preliminary efficacy (prevention of myelosuppression) of Trilaciclib. The second part is a randomized double-blind, placebo-controlled efficacy validation study, and approximately 80 patients with ES-SCLC will be enrolled in Part II, stratified by 1st line vs 2nd/3rd line ES-SCLC, ECOG PS (0-1 vs 2), and presence vs absence of brain metastases, and randomized in a 1:1 ratio to Trilaciclib and placebo, in which patients with 1st line ES-SCLC receive Trilaciclib/placebo combined with EC regimen (Trilaciclib-EC group and placebo-EC group), and patients with 2nd/3rd line ES-SCLC receive Trilaciclib/placebo combined with topotecan (Trilaciclib-TPT group and placeboTPT group), and the efficacy of Trilaciclib (prevention of myelosuppression) will be evaluated with duration of severe neutropenia (DSN) in Cycle 1 as the primary endpoint. The planned dose of Trilaciclib is 240 mg/m2. If the safety data from the first part of the study suggest that the dose of Trilaciclib needs to be adjusted, 12 additional patients (6 patients each for 1st line ES-SCLC and 2nd/3rd line ESSCLC) will be enrolled in the first part of the study to explore the PK and safety of Trilaciclib 200 mg/m2. The study process includes screening period, treatment period, safety followup and survival follow-up.

The end of the study was defined as death in 75% of subjects, or 12 months after the last subject was enrolled, or the sponsor decided to terminate the study, whichever came first.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, male or female;
2. Histologically or cytologically confirmed extensive stage small cell lung cancer (ES-SCLC):

   * Patients scheduled to receive carboplatin plus etoposide regimen: no prior systemic therapy (eg, chemotherapy or combined with immunotherapy);
   * Patients scheduled to receive topotecan regimen: previously received 1/2 lines of chemotherapy or combined immunotherapy but not topotecan.
3. Presence of at least one radiation-naïve measurable lesion according to RECIST 1.1 criteria;
4. Hemoglobin ≥ 90 g/L;
5. Neutrophil count ≥ 1.5 × 10^9/L;
6. Platelet count ≥ 100 × 10^9/L;
7. Creatinine ≤ 15 mg/L or creatinine clearance (CrCl) ≥ 60 mL/min (Cockcroft-Gault formula);
8. Total bilirubin ≤ 1.5 × upper limit of normal (ULN);
9. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN or ≤ 5 × ULN (for patients with liver metastases);
10. Albumin ≥ 30 g/L;
11. ECOG PS score 0 - 2;
12. Expected survival time ≥ 3 months;
13. Contraception:

    Females: All females of childbearing potential must have a negative serum pregnancy test at screening and must use reliable contraception from signing of informed consent through 3 months after the last dose; Male: Female partners of childbearing potential must use reliable contraception from signing the informed consent until 3 months after the last dose;
14. Understand and sign informed consent

Exclusion Criteria:

1. Symptomatic brain metastases requiring local radiotherapy or hormonal therapy;
2. History of other malignancies, with the following exceptions: (1) clinically cured cutaneous basal cell or squamous cell tumors; (2) cured a) cervical cancer, b) prostate cancer, c) superficial bladder cancer; or (3) other solid tumors with a clinical cure time of more than 3 years;
3. Uncontrolled ischemic heart disease or clinically significant congestive heart failure (NYHA Class III or IV);
4. Stroke or cardiovascular or cerebrovascular event within 6 months prior to enrollment;
5. Severe active infection;
6. Psychological or other social factors causing insufficient trial compliance;
7. Other uncontrolled serious chronic diseases or conditions that, in the opinion of the investigator, would make participation in the trial inappropriate;
8. Known HIV infection, active hepatitis B (defined as positive HBV DNA), and hepatitis C (positive HCV RNA);
9. Radiation therapy within 2 weeks prior to enrollment;
10. Patients who have received cytotoxic drug therapy or investigational drug therapy within 4 weeks before enrollment, or non-cytotoxic anti-tumor drug therapy within 2 weeks;
11. Subjects in the first part of the study should not take strong or moderate inducers of CYP3A4 concomitantly within 4 weeks before taking the study drug, and strong inhibitors of CYP3A4 concomitantly within 2 weeks before taking the study drug;
12. Toxicity from prior anticancer therapy has not recovered to Grade 0 or 1 (except alopecia);
13. Hypersensitivity to the study drug (Trilaciclib, etoposide, carboplatin, topotecan) or components thereof;
14. Persons who are unable to act independently due to legal restriction or legal sense;
15. Pregnant or lactating women;
16. Not suitable for participating in this study in the investigator 's opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 95 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ying Cheng, Doctor, Principal Investigator — Jilin Provincial Cancer Hospital
Locations (1):
- Jilin Cancer Hopspital, Changchun, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For Part 1, participants were recruited based on physician referral at 4 academic medical centers ，and the first participant was enrolled on May 25, 2021 and the last participant was enrolled in July 20 2021. For Part 2, participants were recruited based on physician referral at 20 academic medical centers ，and the first participant was enrolled in August 20, 2021 and the last participant was enrolled in December 1 2021.
Pre-assignment Details: For Part 1, of 14 enrolled participants, 12 met inclusion criteria and were treated with trilaicilib plus chemotherapy. For Part 2, of 105 enrolled participants, 83 met inclusion criteria and were randomized to treatment.
Groups:
- Part I ( Safety run-in and PK Evaluation); Trilaciclib Group: 12 patients( 6 patients are first line, 6 patients are second or third line) recieved Trilaciclib(240mg/m^2) plus chemotherapy.
  Patients with first line ES-SCLC received up to 6 cycles of Trilaciclib combined with carboplatin and etoposide or continued treatment until disease progression, intolerability, withdrawal of consent, or investigator termination, whichever came first; patients with second or third line ES-SCLC received Trilaciclib combined with topotecan until disease progression, intolerability, withdrawal of consent, or investigator termination of treatment, whichever came first.
  Carboplatin - administered on Day 1 of each 21-day cycle at a target AUC of 5 (maximum dose 750 mg calculated according to Calvert formula) over 30 min by intravenous infusion; etoposide - administered on Days 1, 2, and 3 of each 21-day cycle at 100 mg/m^2 over 60 min by intravenous infusion; topotecan - administered on Days 1-5 of each 21-day cycle at 1.25 mg/m^2 over 30 min by intravenous infusion.
- Part II ( Randomized Double-blind, Placebo-controlled ), Trilaciclib Group: 41 patients received trilaciclib(240mg/m^2) plus chemotherapy Patients with first line ES-SCLC received up to 6 cycles of Trilaciclib combined with carboplatin and etoposide or continued treatment until disease progression, intolerability, withdrawal of consent, or investigator termination, whichever came first; patients with second or third line ES-SCLC received Trilaciclib combined with topotecan until disease progression, intolerability, withdrawal of consent, or investigator termination of treatment, whichever came first.
  Carboplatin - administered on Day 1 of each 21-day cycle at a target AUC of 5 (maximum dose 750 mg calculated according to Calvert formula) over 30 min by intravenous infusion; etoposide - administered on Days 1, 2, and 3 of each 21-day cycle at 100 mg/m^2 over 60 min by intravenous infusion; topotecan - administered on Days 1-5 of each 21-day cycle at 1.25 mg/m^2 over 30 min by intravenous infusion.
- Part II ( Randomized Double-blind, Placebo-controlled ), Placebo Group: 42 patients received placebo plus chemotherapy Patients with first line ES-SCLC received up to 6 cycles of placebo combined with carboplatin and etoposide or continued treatment until disease progression, intolerability, withdrawal of consent, or investigator termination, whichever came first; patients with second or third line ES-SCLC received placebo combined with topotecan until disease progression, intolerability, withdrawal of consent, or investigator termination of treatment, whichever came first.
  Carboplatin - administered on Day 1 of each 21-day cycle at a target AUC of 5 (maximum dose 750 mg calculated according to Calvert formula) over 30 min by intravenous infusion; etoposide - administered on Days 1, 2, and 3 of each 21-day cycle at 100 mg/m^2 over 60 min by intravenous infusion; topotecan - administered on Days 1-5 of each 21-day cycle at 1.25 mg/m^2 over 30 min by intravenous infusion.
Period: Overall Study
Arm/Group | Part I ( Safety run-in and PK Evaluation); Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Placebo Group
Started | 12 | 41 | 42
Completed | 12 | 41 | 42
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part I ( Safety run-in and PK Evaluation); Trilaciclib Group: 12 patients( 6 patients are first line, 6 patients are second or third line) recieved Trilaciclib(240mg/m^2) plus chemotherapy.
  Patients with first line ES-SCLC received up to 6 cycles of Trilaciclib combined with carboplatin and etoposide or continued treatment until disease progression, intolerability, withdrawal of consent, or investigator termination, whichever came first; patients with second or third line ES-SCLC received Trilaciclib combined with topotecan until disease progression, intolerability, withdrawal of consent, or investigator termination of treatment, whichever came first.
- Part II ( Randomized Double-blind, Placebo-controlled ), Trilaciclib Group: 41 patients received trilaciclib(240mg/m^2) plus chemotherapy Patients with first line ES-SCLC received up to 6 cycles of Trilaciclib combined with carboplatin and etoposide or continued treatment until disease progression, intolerability, withdrawal of consent, or investigator termination, whichever came first; patients with second or third line ES-SCLC received Trilaciclib combined with topotecan until disease progression, intolerability, withdrawal of consent, or investigator termination of treatment, whichever came first.
- Part II ( Randomized Double-blind, Placebo-controlled ), Placebo Group: 42 patients received placebo plus chemotherapy Patients with first line ES-SCLC received up to 6 cycles of placebo combined with carboplatin and etoposide or continued treatment until disease progression, intolerability, withdrawal of consent, or investigator termination, whichever came first; patients with second or third line ES-SCLC received placebo combined with topotecan until disease progression, intolerability, withdrawal of consent, or investigator termination of treatment, whichever came first.
- Total: Total of all reporting groups
Arm/Group | Part I ( Safety run-in and PK Evaluation); Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Placebo Group | Total
Number analyzed (Participants) | 12 | 41 | 42 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (7.06) | 62.0 (7.78) | 59.4 (8.71) | 60.7 (8.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 33 | 35 | 77
  Male | 3 | 8 | 7 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 12 | 41 | 42 | 95
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 12 | 41 | 42 | 95
Brain metastases at baseline [Number; unit: participants] | 5 | 13 | 16 | 34

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero Extrapolated to Infinity(AUC0-inf) for Part 1
Description: AUC0-inf of trilaciclib in plasma was determined from individual concentration-time data by non-compartmental analysis methods. The actual sampling times in relation to dosing were used.
Time Frame: Day1 and Day 3( or Day 5) of Cycle 1 for a 21-day cycle
Population: PK Analysis Set (PKS): All patients who received at least one dose of the study drug and had at least one valid concentration data of the tested components after drug administration. Pharmacokinetic analyses will be based on the PKS set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Part I ( Safety run-in and PK Evaluation); Trilaciclib Group, First Line ES-SCLC: Trilaciclib 240 mg/m^2 in patients with first line ES-SCLC receiving carboplatin plus etoposide chemotherapy
- Part I ( Safety run-in and PK Evaluation); Trilaciclib Group, Second or Third Line ES-SCLC: Trilaciclib 240 mg/m^2 in patients in patients with second or third line ES-SCLC receiving topotecan chemotherapy
Arm/Group | Part I ( Safety run-in and PK Evaluation); Trilaciclib Group, First Line ES-SCLC | Part I ( Safety run-in and PK Evaluation); Trilaciclib Group, Second or Third Line ES-SCLC
Number analyzed (Participants) | 6 | 6
h*ng/mL
  Day 1 Cycle 1 | 2200 (14.5) | 2598 (23.5)
  first line: Day 3 Cycle 1 Second or third line: Day 5 Cycle 1 | 2878 (38.6) | 2675 (22.0)

2. Primary Outcome: Duration of Severe Neutropenia in Cycle 1 (DSN)
Description: DSN in Cycle 1 was defined as the number of days from the date of the first ANC value < 0.5 x 10^9/L in Cycle 1 to the date of the first ANC value ≥ 0.5 x 10^9/L. The date of the first ANC value ≥ 0.5 x 10^9/L should meet the following requirements: (1) occurred after the ANC value was < 0.5 x 10^9/L, and (2) there were no other ANC values < 0.5 x 10^9/L between this date and the end of Cycle 1 (otherwise, if this patient entered Cycle 2, it was counted as Day 1 of Cycle 2). DSN in Cycle 1 was scored as 0 if the patient did not experience any SN during Cycle 1.
Time Frame: At the end of Cycle 1 (each cycle is 21 days)
Population: The FAS included all enrolled patients who received at least one dose of study drug according to the intention-to-treat (ITT) principle.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Part I ( Safety run-in and PK Evaluation); Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Placebo Group
Number analyzed (Participants) | 12 | 41 | 42
Days | 0.7 (2.31) | 0 (1.7) | 2 (3.0)
Statistical Analysis 1: Comparison: Part II ( Randomized Double-blind, Placebo-controlled ), Trilaciclib Group vs Part II ( Randomized Double-blind, Placebo-controlled ), Placebo Group; 70 subjects (35 per group) provided approximately 95% power at the test level of α = 0.05 (2-sided) .Assuming a dropout rate of approximately 12%, the sample size for Part II was 80 subjects (40 per group); Test type: Superiority; p = 0.0003, non-parametric ANCOVA

3. Primary Outcome: Maximum Observed Plasma Concentration(Cmax) of Trilaciclib for Part 1
Description: Cmax of trilaciclib in plasma was determined from individual concentration-time data by non-compartmental analysis methods. The actual sampling times in relation to dosing were used. For estimation of Cmax, a concentration that was below the limit of quantification (BLQ) was assigned a value of zero if it occurred in a profile before the first measurable concentration. If a BLQ value occurred after a measurable concentration in a profile, and was followed by a value above the lower limit of quantification, then the BLQ was treated as missing data. If a BLQ value occurred at the end of the collection interval (after the last quantifiable concentration) it was treated as missing data. If two BLQ values occurred in succession after Cmax, the profile was deemed to have terminated at the first BLQ value and any subsequent concentrations were omitted.
Time Frame: Day1 and Day 3( or Day 5) of Cycle 1 for a 21-day cycle
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part I ( Safety run-in and PK Evaluation); Trilaciclib Group, First Line ES-SCLC | Part I ( Safety run-in and PK Evaluation); Trilaciclib Group, Second or Third Line ES-SCLC
Number analyzed (Participants) | 6 | 6
ng/mL
  Day 1 Cycle 1 | 1007 (18.8) | 918 (46.7)
  First line: Day 3 Cycle 1 Second or third line: Day 5 Cycle 1 | 893 (36.2) | 776 (29.9)

4. Secondary Outcome: Occurrence of Severe Neutropenia (SN)
Description: Severe (Grade 4) neutropenia was defined as at least 1 ANC value <0.5 × 10^9/L during the treatment period.
Time Frame: From date of randomization , 21 day treatment cycle to the end of the treatment until (if earlier) disease progression, start of subsequent anticancer treatment, withdrawal of informed consent, or death, acessed up to a maximum of 12 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part I ( Safety run-in and PK Evaluation); Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Placebo Group
Number analyzed (Participants) | 12 | 41 | 42
Participants | 2 | 4 | 20

5. Secondary Outcome: Occurrence of Red Blood Cell Transfusion (on/After Week 5)
Description: The occurrence of RBC transfusions was defined as at least 1 cycle with RBC transfusion during the treatment period. For the treatment period, the total number of RBC transfusions was the number of cycles with RBC transfusions.
Time Frame: From week 5 to the end of the treatment until (if earlier) disease progression, start of subsequent anticancer treatment, withdrawal of informed consent, or death, acessed up to a maximum of 12 months
Population: The FAS included all randomized patients who received at least one dose of study drug according to the intention-to-treat (ITT) principle.
Measure: Count of Participants; unit: Participants
Arm/Group | Part I ( Safety run-in and PK Evaluation); Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Placebo Group
Number analyzed (Participants) | 12 | 41 | 42
Participants | 0 | 2 | 2

6. Secondary Outcome: Granulocyte Colony Stimulating Factor (G-CSF) Use Rate
Description: Administration of G-CSF was collected with concomitant medications, which were coded using World Health Organization Drug Dictionary (WHO-DD) . A cycle where G-CSF was administered concurrently was identified by comparing the start and stop dates of each administration of G-CSF to the start of cycle and end of cycle. The occurrence of G-CSF administrations was defined as at least 1 cycle with G-CSF administrations during the treatment period. For the treatment period, the total number of G-CSF administrations was the number of cycles with G-CSF administrations.
Time Frame: as for outcome 4
Population: The FAS included all randomized patients who received at least 1 dose of study drug according to the intention-to-treat (ITT) principle.
Measure: Count of Participants; unit: Participants
Arm/Group | Part I ( Safety run-in and PK Evaluation); Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Placebo Group
Number analyzed (Participants) | 12 | 41 | 42
Participants | 4 | 28 | 29

7. Secondary Outcome: Composite Endpoints-major Hematologic AEs (Anyone of the Followings): All-cause Hospitalization; All-cause Dose Reductions; Febrile Neutropenia; SN Prolongation (Lasting > 5 Days); Red Blood Cell (RBC) Transfusions Were Performed on/After Week 5.
Description: MAHE was a composite endpoint incorporating the measurement of several clinically meaningful aspects of myelopreservation into a single endpoint. The individual components for MAHE were hospitalization for a hematologic event, febrile neutropenia, death related to treatment, dose delay/reduction due to ANC or platelet counts, prolonged severe neutropenia (duration >5 days), RBC transfusion (actual or eligible) and platelet transfusion (actual or eligible).
  Event rate per week， calculated as the total number of events divided by duration of in weeks.
Time Frame: as for outcome 4
Population: as for outcome 6
Measure: Number; unit: events per week
Arm/Group | Part I ( Safety run-in and PK Evaluation); Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Placebo Group
Number analyzed (Participants) | 12 | 41 | 42
events per week | 0.033 | 0.040 | 0.077

8. Secondary Outcome: Occurrence of Grade 3 and 4 Hematological Toxicities
Description: Occurrence of Grade 3 and 4 hematological toxicities was defined according to CTCAE 5.0 during the treatment period.
Time Frame: as for outcome 4
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Part I ( Safety run-in and PK Evaluation); Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Placebo Group
Number analyzed (Participants) | 12 | 41 | 42
Participants | 6 | 24 | 38

9. Secondary Outcome: Erythropoiesis Stimulating Agent (ESA) Use Rate
Description: Administration of ESA was collected with concomitant medications, which were coded using WHO-DD . A cycle where an ESA was administered concurrently was identified by comparing the start and stop dates of each administration of an ESA to the start of cycle and end of cycle. The occurrence of ESA administration was at least 1 cycle with an ESA administration during the treatment period. For the treatment period, the total number of ESA administrations was the number of cycles with ESA administrations.
Time Frame: as for outcome 4
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Part I ( Safety run-in and PK Evaluation); Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Placebo Group
Number analyzed (Participants) | 12 | 41 | 42
Participants | 1 | 6 | 8

10. Secondary Outcome: Recombinant Human Interleukin-11 Use Rate
Description: Administration of interleukin-11 was collected with concomitant medications, which were coded using WHO-DD Version. A cycle where interleukin-11 was administered concurrently was identified by comparing the start and stop dates of each administration of interleukin-11 to the start of cycle and end of cycle. The occurrence of interleukin-11 administration was at least 1 cycle with interleukin-11 administration during the treatment period.
Time Frame: as for outcome 4
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Part I ( Safety run-in and PK Evaluation); Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Placebo Group
Number analyzed (Participants) | 12 | 41 | 42
Participants | 2 | 12 | 11

11. Secondary Outcome: Thrombopoietin (TPO) Use Rate
Description: Administration of TPO was collected with concomitant medications, which were coded using WHO-DD Version. A cycle where TPO was administered concurrently was identified by comparing the start and stop dates of each administration of TPO to the start of cycle and end of cycle. The occurrence of TPO administration was at least 1 cycle with TPO administration during the treatment period.
Time Frame: as for outcome 4
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Part I ( Safety run-in and PK Evaluation); Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Placebo Group
Number analyzed (Participants) | 12 | 41 | 42
Participants | 4 | 10 | 10

12. Secondary Outcome: Occurrence of Intravenous or Oral Antibiotic Administration
Description: Administration of intravenous or oral antibiotic was collected with concomitant medications, which were coded using WHO-DD Version. A cycle where intravenous or oral antibiotic was administered concurrently was identified by comparing the start and stop dates of each administration of intravenous or oral antibiotic to the start of cycle and end of cycle. The occurrence of intravenous or oral antibiotic administration was at least 1 cycle with intravenous or oral antibiotic administration during the treatment period.
Time Frame: as for outcome 4
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Part I ( Safety run-in and PK Evaluation); Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Placebo Group
Number analyzed (Participants) | 12 | 41 | 42
Participants | 3 | 11 | 13

13. Secondary Outcome: Occurrence of Infectious Serious Adverse Events
Description: SAEs were defined as any untoward medical occurrence that at any dose resulted in death, was life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity or was a congenital anomaly/birth defect. An infectious SAE was a serious event in the Medical Dictionary for Regulatory Activities (MedDRA) system organ class "infections and infestations" and a preferred term of anal abscess, bacteraemia, bronchitis, candida infection, chronic sinusitis, conjunctivitis, infection, influenza, nasopharyngitis, oral candidiasis, oral herpes, pharyngitis streptococcal, pneumonia, pneumonia bacterial, respiratory tract infection, sepsis, skin infection, upper respiratory tract infection, urinary tract infection, urosepsis or viral upper respiratory tract infection.
Time Frame: as for outcome 4
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Part I ( Safety run-in and PK Evaluation); Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Placebo Group
Number analyzed (Participants) | 12 | 41 | 42
Participants | 0 | 1 | 0

14. Secondary Outcome: Occurrence of Lung Infection SAEs
Description: SAEs were defined as any untoward medical occurrence that at any dose resulted in death, was life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity or was a congenital anomaly/birth defect. A lung infection SAE was a serious event in the MedDRA system organ class "infections and infestations" and a preferred term of bronchitis, influenza, pneumonia, pneumonia bacterial, respiratory tract infection, upper respiratory tract infection or viral upper respiratory tract infection.
Time Frame: as for outcome 4
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Part I ( Safety run-in and PK Evaluation); Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Placebo Group
Number analyzed (Participants) | 12 | 41 | 42
Participants | 0 | 1 | 0

15. Secondary Outcome: Occurrence of Febrile Neutropenia
Description: Each febrile neutropenia event (as defined by Common Terminology Criteria for Adverse Events [CTCAE]) was captured as an AE. The occurrence of febrile neutropenia was defined as at least 1 febrile neutropenia event during the treatment period. For the treatment period, the total number of febrile neutropenia events was the number of febrile neutropenia events with a unique start date.
Time Frame: as for outcome 4
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Part I ( Safety run-in and PK Evaluation); Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Placebo Group
Number analyzed (Participants) | 12 | 41 | 42
Participants | 1 | 1 | 7

16. Secondary Outcome: Occurrence of Platelet Transfusion
Description: The occurrence of platelet transfusions was defined as at least 1 cycle with platelet transfusion during the treatment period. For the treatment period, the total number of platelet transfusions was the number of cycles with platelet transfusions.
Time Frame: as for outcome 4
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Part I ( Safety run-in and PK Evaluation); Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Placebo Group
Number analyzed (Participants) | 12 | 41 | 42
Participants | 0 | 3 | 4

17. Secondary Outcome: Objective Tumor Response Rate (ORR)
Description: ORR was performed based on the Response Evaluation Analysis Set (RES). Based on the assessments at each visit, the number and percentage of patients with best response of CR, PR, SD, PD and NE will be summarized by treatment group when CR/PR confirmation is not required and CR/PR confirmation is required, respectively . In particular, SD BOR requires at least 35 days or more after enrollment.ORR was calculated based on the number of patients with best response of CR or PR.
Time Frame: From date of randomization , 21 day treatment cycle to the end of the treatment until (if earlier) disease progression, start of subsequent anticancer treatment, withdrawal of informed consent, or death, acessed up to a maximum of 18 months
Population: Response Evaluable Analysis Set (RES): all patients who took at least one dose of study drug, had measurable disease at baseline, and completed at least one post-treatment tumor imaging assessment. This analysis set was used for the analysis of anti-tumor efficacy endpoints related to tumor RECIST1.1 assessment.
  efficacy endpoints related to tumor RECIST1.1 assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part I ( Safety run-in and PK Evaluation); Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Placebo Group
Number analyzed (Participants) | 9 | 38 | 38
Participants | 2 | 17 | 15

18. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was performed based on the Response Evaluation Analysis Set (RES). Based on the assessments at each visit, the number and percentage of patients with best response of CR, PR, SD, PD and NE will be summarized by treatment group when CR/PR confirmation is not required and CR/PR confirmation is required, respectively . In particular, SD BOR requires at least 35 days or more after enrollment. DCR was calculated based on the number of patients with best response of CR PR or SD.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Part I ( Safety run-in and PK Evaluation); Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Placebo Group
Number analyzed (Participants) | 9 | 38 | 38
Participants | 8 | 32 | 31

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from the time of informed consent through the end of the safety follow-up period, initiation of new antineoplastic therapy, or withdrawal from the study, whichever came first, acessed up to a maximum of 18 months
Arm/Group | Part I ( Safety run-in and PK Evaluation); Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Trilaciclib Group | Part II ( Randomized Double-blind, Placebo-controlled ), Placebo Group
All-Cause Mortality (participants affected / at risk) | 6/12 | 22/41 | 28/42
Serious Adverse Events (participants affected / at risk) | 4/12 | 12/41 | 15/42
Other Adverse Events (participants affected / at risk) | 12/12 | 41/41 | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part I ( Safety run-in and PK Evaluation); Trilaciclib Group (N=12) | Part II ( Randomized Double-blind, Placebo-controlled ), Trilaciclib Group (N=41) | Part II ( Randomized Double-blind, Placebo-controlled ), Placebo Group (N=42)
Neutrophil count decreased (Investigations) | 1 | 2 | 5
Platelet count decreased (Investigations) | 1 | 5 | 6
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 3
Pyrexia (General disorders) | 0 | 1 | 0
Oxygen saturation decreased (Investigations) | 1 | 0 | 0
acute cardiac failure (Cardiac disorders) | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 2
Disease progression (General disorders) | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part I ( Safety run-in and PK Evaluation); Trilaciclib Group (N=12) | Part II ( Randomized Double-blind, Placebo-controlled ), Trilaciclib Group (N=41) | Part II ( Randomized Double-blind, Placebo-controlled ), Placebo Group (N=42)
Neutrophil count decreased (Investigations) | 7 | 33 | 40
Platelet count decreased (Investigations) | 6 | 28 | 34
White blood cell count decreased (Investigations) | 7 | 32 | 42
Alanine aminotransferase increased (Investigations) | 5 | 11 | 12
Aspartate aminotransferase increased (Investigations) | 4 | 8 | 10
Gamma-glutamyltransferase increased (Investigations) | 2 | 12 | 10
Blood alkaline phosphatase increased (Investigations) | 2 | 7 | 5
Lymphocyte count decreased (Investigations) | 4 | 8 | 11
Blood bilirubin increased (Investigations) | 0 | 3 | 6
Blood lactate dehydrogenase increased (Investigations) | 2 | 4 | 5
Nausea (Gastrointestinal disorders) | 5 | 13 | 14
Constipation (Gastrointestinal disorders) | 0 | 13 | 18
Vomiting (Gastrointestinal disorders) | 4 | 5 | 8
Anaemia (Blood and lymphatic system disorders) | 8 | 28 | 35
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 5 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 8 | 11
decreased appetite (Metabolism and nutrition disorders) | 5 | 6 | 13
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 5 | 4
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 7 | 12 | 9
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 4 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 8 | 12
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 7 | 10
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 7 | 12
Weight decreased (Investigations) | 0 | 6 | 2
Asthenia (General disorders) | 3 | 3 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 3 | 5
pyrexia (General disorders) | 0 | 7 | 6
Insomnia (Psychiatric disorders) | 1 | 5 | 5
sinus tachycardia (Cardiac disorders) | 0 | 4 | 5
proteinuria (Renal and urinary disorders) | 2 | 4 | 2
Hematuria (Renal and urinary disorders) | 0 | 4 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 3 | 6
cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 6
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 3 | 3
hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 3 | 3
back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3
Increased serum creatinine (Renal and urinary disorders) | 3 | 2 | 1
urinary tract infection (Infections and infestations) | 2 | 3 | 0
Chest discomfort (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Phlebitis (Vascular disorders) | 1 | 3 | 0
Hyperlipidemia (Metabolism and nutrition disorders) | 0 | 3 | 3
Headache (Nervous system disorders) | 0 | 2 | 5
hypophosphatemia (Metabolism and nutrition disorders) | 1 | 2 | 3
Dizziness (Nervous system disorders) | 1 | 2 | 3
Pain in limb (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 1 | 1 | 0
Tricuspid valve insufficiency (Cardiac disorders) | 1 | 0 | 0
Aortic valve insufficiency (Cardiac disorders) | 1 | 0 | 0
Mitral valve insufficiency (Cardiac disorders) | 1 | 0 | 0
Weight increased (Investigations) | 1 | 2 | 2
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 1
Urine occult blood positive (Investigations) | 1 | 2 | 0
Hypoaesthesia (General disorders) | 1 | 0 | 1
Injection site pain (General disorders) | 1 | 0 | 0
Decreased range of motion (General disorders) | 1 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0
Fibrin D-dimer increased (Investigations) | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Troponin T increased (Investigations) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2
Blood urea increased (Investigations) | 1 | 2 | 1
Blood myoglobin increased (Investigations) | 1 | 0 | 0
Blood creatine phosphokinase MB increased (Investigations) | 1 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 2 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 0
Embolism (Vascular disorders) | 1 | 2 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 2 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/85/NCT04902885/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-16): https://cdn.clinicaltrials.gov/large-docs/85/NCT04902885/SAP_001.pdf